CLINICAL TRIAL: NCT01647594
Title: Qualitative Assessment and Pilot Study for Young Women's Intervention
Brief Title: Pilot Study for Young Women's Intervention
Acronym: YWI Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-390
Record Dates: First submitted 2011-10-26; First posted 2012-07-23 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Young women; Fertility; Physical activity; Survivorship
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young Women's Intervention (YWI) (Active Comparator)
  Interventions: Behavioral: YWI
- Physical Activity Intervention (PAI) (Active Comparator)
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: YWI — The YWI consists of print and web-based materials. Content for this group will include detailed information about issues facing young women with breast cancer, risks, discussion points and and resources. The following domains will be addressed: health/medical issues (i.e., side effects, breast cancer recurrence, long-term risks, genetic issues), psychosocial issues (coping, relationship and family concerns), beauty/body image, sexual functioning, fertility concerns, and work/school issues.
  Arms: Young Women's Intervention (YWI)
Behavioral: Physical Activity — The PAI serves as the control group. This intervention consists of print and web-based materials, the content of which includes detailed information about the benefits of exercise in breast cancer survivors and discussion points, available options and resources to enhance physical activity after diagnosis.
  Arms: Physical Activity Intervention (PAI)

SUMMARY:
This is a pilot study, which will inform a larger study to evaluate the Young Women's Intervention (YWI). The goal of this research is to develop, implement and test a refined exportable and sustainable education and support intervention for young women with breast cancer and their oncology providers. This pilot study will test the feasibility of the Young Women's Intervention (YWI) as well as a Physical Activity Intervention (PAI) at four unique sites. In addition, it will include a qualitative assessment, through focus groups and key informant interviews, of concerns facing young women with breast cancer. The investigators aim to use the findings from this pilot study to inform a larger future Young Women's Intervention (YWI) study where the YWI intervention will be compared to a Physical Activity Intervention (PAI).

DETAILED DESCRIPTION:
Breast cancer in young women is a not a common disease, yet over 12,000 women under 40 are diagnosed with invasive breast cancer yearly in the United States alone and an additional 2,000 are diagnosed with noninvasive disease. Breast cancer is the leading cause of cancer-related deaths in women under 40, and survival rates for young women with breast cancer are lower than for their older counterparts. Further, in addition to being at higher risk of dying from breast cancer, despite often receiving more aggressive therapy, young women are at higher risk of distress both at diagnosis and in follow-up. Young women often have multiple roles and responsibilities that are harder to adjust to or get others to take on (e.g., parenting of young children, completing education, or building a career). Many young women are interested in having biologic children following treatment and are concerned about their future fertility. They also have an increased risk of harboring a genetic risk factor for breast cancer. Finally, in contrast to older women with breast cancer, who represent the majority of women with the disease, young women often feel isolated and lacking information, and they sometimes are concerned that their doctors are unsure of how to treat them. Distress may be confounded by lack of information on some of the risks they face, lack of provider awareness, information, and resources to address young women's concerns, and lack of peer support. These issues may contribute to the greater psychosocial distress seen in younger women at both diagnosis and in follow-up compared with older women. Thus, attention to these issues in younger women is warranted. Yet, research has revealed that needs of young women are not being met.

The primary goals of this study are to:

1. conduct a qualitative assessment, through focus groups and key informant interviews, of concerns facing young women with breast cancer;
2. evaluate materials developed to provide young women newly diagnosed with breast cancer information and resources regarding their unique concerns or physical activity through focus groups and a pilot study;
3. conduct a pilot study of the Young Women's Intervention (YWI) as well as a Physical Activity Intervention (PAI) at 4 unique sites (3 will use the YWI and 2 will use the PAI- DFCI will pilot both interventions, one following the other) to evaluate the process for the intervention as well as to pilot surveys.

We aim to use the findings from the focus groups, key informant interviews and pilot study to inform the larger future Young Women's Intervention (YWI) study where the YWI arm will be compared to a Physical Activity Intervention (PAI). We plan to develop, implement and test a refined exportable and sustainable education and support intervention for young women with breast cancer and their oncology providers. First, we want to conduct focus groups and key informant interviews aiming to qualitatively assess the following domains: health/medical issues (i.e. side effects, breast cancer recurrence, long-term risks, genetic issues), psychosocial issues (coping, relationship and family concerns), beauty/body image, sexual functioning, fertility concerns, and work/school issues. In addition, the focus groups will be used to review the study materials and provide constructive feedback. In order to get a more diverse view of young women's concerns, we will conduct key informant interviews by telephone with young women with a history of breast cancer recruited from various regions of the country.

Information gained through the focus groups, key informant interviews and pilot of the intervention at four diverse practices will help us discover and resolve issues related to: administering the baseline survey, follow-up survey and provider survey; ensuring that the adapted intervention meets patient and provider needs, and evaluation the implementation process. When evaluating the patient surveys, investigators will assess issues that may have posed a barrier to patients' comprehension of study questions, such as the use of jargon or difficult vocabulary. In addition to piloting patient and provider surveys for material content, we will evaluate the intervention for feasibility of recruitment and implementation. We will refine materials and methods based on our pilot experience.

Collectively, results from the qualitative assessment and pilot will help finalize materials and surveys as well the methods of the study for a planned multi-site intervention study (YWI) funded by ASCO with support from Susan G. Komen for the Cure. A detailed plan of the parent study intervention will be submitted to the IRB upon completion of the focus groups, key informant interviews and pilot study described above.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write English
* Age 18-42 at time of diagnosis
* Within 4 years of stage I-III invasive breast cancer diagnosis
* No known recurrence or metastatic disease
* Subject can be under active treatment at the time of study participation

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of intervention materials in addressing the unique issues facing young women with breast cancer | 1 year
  Through focus groups and a pilot study, we will evaluate materials developed to provide young women newly diagnosed with breast cancer information and resources regarding their unique concerns or physical activity.
Evaluate process of intervention | 1 year
  This pilot study is being conducted at 4 unique sites to assess the feasibility of recruitment and implementation, as well as to pilot the surveys.
Qualitative assessment of concerns facing young women with breast cancer | 1 year
  The qualitative assessment will entail moderated in-person focus groups and key informant phone interviews, both of which will explore issues concerning young women with newly-diagnosed breast cancer. The following domains will be assessed: health/medical issues (i.e. side effects, breast cancer recurrence, long-term risks, genetic issues), psychosocial issues (coping, relationship and family concerns), beauty/body image, sexual functioning, fertility concerns, and work/school issues.

SECONDARY OUTCOMES:
Efficacy of materials for helping providers improve cancer treatment for young women with breast cancer | Baseline, and about one week later
  During the pilot intervention, we will pilot two patient surveys and one provider survey for material content and feedback on the intervention materials.

CONTACTS AND LOCATIONS:
Overall Officials: Ann H. Partridge, M.D., M.P.H., Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Eastern Maine Medical Center, Brewer, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Texas Oncology Cancer Center, Houston, Texas